CLINICAL TRIAL: NCT03039101
Title: Double Blind Study of Leukotriene Antagonism in the Nasal Recruitment of CD49d Expressing Neutrophils in Atopic Subjects
Brief Title: Leukotriene Antagonism in Recruitment of CD49d Expressing Neutrophils in Atopic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mitchell Grayson (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Mitchell Grayson, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB16-00842; R01HL087778 (NIH)
Record Dates: First submitted 2017-01-26; First posted 2017-02-01 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Nasal Allergy
Keywords: allergen; neutrophils; allergy
MeSH Terms: conditions — Hypersensitivity | interventions — Nasal Lavage; montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Montelukast (Experimental): Subjects take 1 montelukast 10mg tablet orally, daily and effect on nasal allergen challenge (based on results of epicutaneous skin testing) induced recruitment of cd49d neutrophils in the peripheral blood and nasal lavage determined at 1 week
  Interventions: Procedure: Nasal lavage; Procedure: Nasal allergen challenge; Procedure: Epicutaneous skin testing; Procedure: Peripheral blood; Drug: Montelukast 10Mg Tablet
- Placebo (Placebo Comparator): Subjects take 1 placebo oral pill, daily and effect on nasal allergen challenge (based on results of epicutaneous skin testing) induced recruitment of cd49d neutrophils in the peripheral blood and nasal lavage determined at 1 week.
  Interventions: Procedure: Nasal lavage; Procedure: Nasal allergen challenge; Procedure: Peripheral blood; Drug: Placebo Oral Tablet

INTERVENTIONS:
Procedure: Nasal lavage — determine frequency of CD49d expressing neutrophils in the nasal lavage by flow cytometry
Procedure: Nasal allergen challenge — A small amount of allergen extract will be applied to one naris.
Procedure: Epicutaneous skin testing — Skin testing (prick) to determine allergies.
  Arms: Montelukast
Procedure: Peripheral blood — Peripheral blood draw
Drug: Montelukast 10Mg Tablet — one pill orally, daily, for 1 week
  Other Names: montelukast
  Arms: Montelukast
Drug: Placebo Oral Tablet — one pill orally, daily, for 1 week
  Other Names: placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if the recruitment of a certain cell type (the alpha 4 integrin (CD49d) expressing neutrophil) during a nasal allergen challenge can be inhibited by pretreatment with an FDA approved leukotriene antagonist (montelukast).

DETAILED DESCRIPTION:
Subjects will be consented, undergo skin testing, medical history questionnaires, and randomized to either placebo or montelukast (10 mg). In one week, subjects return, undergo a blood draw, medical history questionnaires, nasal lavage, and nasal allergen challenge (followed by lavage in 6 hours). Subjects will then cross-over to the other study drug. One week later subjects will undergo a blood draw, medical history questionnaires, lavage, allergen challenge, and repeat lavage (after 6 hours).

ELIGIBILITY:
Inclusion Criteria:

* 21 - 65 years of age, inclusive
* A personal history of allergic rhinitis (hayfever) (by self-report)
* At least one positive skin test to cat, dust mite mix, Timothy grass, Bermuda grass, Bluegrass, or Ragweed
* Ability to provide informed consent
* Willingness to undergo epicutaneous skin testing
* Willingness to undergo nasal lavages and nasal allergen challenges
* Willingness to undergo 2 peripheral blood draws (10 cc each)

Exclusion Criteria:

* Use of systemic antihistamine in the past 5 days
* Use of intranasal corticosteroids or intranasal antihistamines currently or in the past 2 weeks
* Use of Montelukast currently or in the past week
* Hypersensitivity or allergy to Montelukast
* Inability to perform/undergo any study procedures
* Pregnancy (by subject report) or breastfeeding
* Confirmed or suspected immunodeficiency
* Persistent asthma, atopic dermatitis, or any other co-morbid disease except for allergic rhinitis
* Any symptoms of asthma in the past 2 weeks (shortness of breath, wheezing, and/or use of albuterol)
* Fever (temperature over 99F) currently or in the past 2 weeks
* Current or previous use of a biologic or investigational agent in the past 6 months
* Current or past suicidal thoughts/attempts

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-07-16 (Actual)

PRIMARY OUTCOMES:
Change in frequency in CD49d+ neutrophils in the nasal lavage post-allergen challenge on placebo versus Montelukast. | 1 month
  The primary outcome will be the change in frequency (as assessed by flow cytometry) in CD49d+ neutrophils in the nasal lavage post-allergen challenge on placebo versus Montelukast.

SECONDARY OUTCOMES:
Change in clinical response following nasal allergen challenge after one week of treatment with Montelukast. | 1 month
  Secondary outcomes will be whether treatment with Montelukast for one week changes the clinical response to nasal allergen challenge (i.e., sneezing, itching, etc.) as documented in the validated Sino Nasal Outcome Test (SNOT)-20 questionnaire.

OTHER OUTCOMES:
Induction of expression of immunoglobulin E (IgE) receptor on dendritic cells following exposure with CD49d+ cells from peripheral blood samples. | 1 month
  An additional outcome will be whether CD49d+ neutrophils from peripheral blood can induce increased expression of the IgE receptor (FceRI) on dendritic cells (also isolated from the peripheral blood).

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell H Grayson, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sigua JA, Buelow B, Cheung DS, Buell E, Hunter D, Klancnik M, Grayson MH. CD49d-expressing neutrophils differentiate atopic from nonatopic individuals. J Allergy Clin Immunol. 2014 Mar;133(3):901-4.e5. doi: 10.1016/j.jaci.2013.09.035. Epub 2013 Dec 18. No abstract available. PMID 24360325
- [Background] Cheung DS, Ehlenbach SJ, Kitchens RT, Riley DA, Thomas LL, Holtzman MJ, Grayson MH. Cutting edge: CD49d+ neutrophils induce FcepsilonRI expression on lung dendritic cells in a mouse model of postviral asthma. J Immunol. 2010 Nov 1;185(9):4983-7. doi: 10.4049/jimmunol.1002456. Epub 2010 Sep 27. PMID 20876348
- [Background] Khan SH, Grayson MH. Cross-linking IgE augments human conventional dendritic cell production of CC chemokine ligand 28. J Allergy Clin Immunol. 2010 Jan;125(1):265-7. doi: 10.1016/j.jaci.2009.09.038. Epub 2009 Dec 4. No abstract available. PMID 19962743
- [Background] Subrata LS, Bizzintino J, Mamessier E, Bosco A, McKenna KL, Wikstrom ME, Goldblatt J, Sly PD, Hales BJ, Thomas WR, Laing IA, LeSouef PN, Holt PG. Interactions between innate antiviral and atopic immunoinflammatory pathways precipitate and sustain asthma exacerbations in children. J Immunol. 2009 Aug 15;183(4):2793-800. doi: 10.4049/jimmunol.0900695. Epub 2009 Jul 20. PMID 19620293
- [Background] Cheung DS, Ehlenbach SJ, Kitchens T, Riley DA, Grayson MH. Development of atopy by severe paramyxoviral infection in a mouse model. Ann Allergy Asthma Immunol. 2010 Dec;105(6):437-443.e1. doi: 10.1016/j.anai.2010.09.010. PMID 21130381
- [Background] Grayson MH, Cheung D, Rohlfing MM, Kitchens R, Spiegel DE, Tucker J, Battaile JT, Alevy Y, Yan L, Agapov E, Kim EY, Holtzman MJ. Induction of high-affinity IgE receptor on lung dendritic cells during viral infection leads to mucous cell metaplasia. J Exp Med. 2007 Oct 29;204(11):2759-69. doi: 10.1084/jem.20070360. Epub 2007 Oct 22. PMID 17954569
- [Background] Sigurs N, Bjarnason R, Sigurbergsson F, Kjellman B, Bjorksten B. Asthma and immunoglobulin E antibodies after respiratory syncytial virus bronchiolitis: a prospective cohort study with matched controls. Pediatrics. 1995 Apr;95(4):500-5. PMID 7700748
- [Result] Sammon LM, Hussain SA, Smith M, Rohlfing M, Santoro JL, Grayson MH. Effect of cysteinyl leukotriene receptor 1 blockade on aeroallergen-induced nasal recruitment of CD49d expressing neutrophils. Ann Allergy Asthma Immunol. 2019 Nov;123(5):508-511.e1. doi: 10.1016/j.anai.2019.08.019. Epub 2019 Sep 3. No abstract available. PMID 31491537